CLINICAL TRIAL: NCT03228173
Title: Iron Deficiency, Depression, and Other Affective Disorders in Female State Fair Attendees
Brief Title: Iron Deficiency in Female State Fair Attendees
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of Hawaii (Other)
Responsible Party: Sponsor
Other Study IDs: State Fair
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Iron Deficiency (Without Anemia)
Keywords: Cognition; Executive functioning; Depression; Affect; adult females
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum from each subject was coded and frozen in a -80 degrees C in a lab at the University of Minnesota
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to examine iron deficiency symptoms and biochemical iron status based on hemoglobin, hematocrit, ferritin, and total iron binding capacity in menstruating females.

DETAILED DESCRIPTION:
Iron deficiency affects nearly 2 billion people globally, and it is among the most common risk factors for disability and death. In its most extreme presentation, it results in anemia, where the RBC count of the individual is markedly low, hindering oxygen transport. Anemia has a remarkable global presence, affecting approximately one third of the world's population. Though there are multiple causes for anemia, the World Health Organization (WHO) estimates that the most common cause for anemia on the planet is iron deficiency. Although findings from the US indicate that iron deficiency is less prevalent than in many other nations, iron deficiency is still a pervasive national public health concern. A study that analyzed the National Health and Nutrition Examination Survey (NHANES) data from 2007-2010 indicated that US children 5 years of age and younger have an anemia incidence of 3.2 percent.

Incidence of depression varies based on diagnostic tools used and categories included, as well as the country, gender, age, and socioeconomic status of individuals. Globally, it is estimated that between 4 and 10 percent of people experience major depressive disorder (MDD) while between 2.5 and 5 percent experience dysthymia, a depression that involves less severe symptoms but has a chronic manifestation. On average, the first onset of depression is 20 years old, though this figure is highly variable. It has consistently been demonstrated that females experience a much higher incidence of depression than males. MDD has repeatedly been reported in females at rates 1.5 to 3 times that of males, and female dysthymia has been reported at 2 times that of males.

The current state of the literature on the connection between mental health and iron status is further muddled by subjective, self-reported assessments and a lack of randomized controlled trials, but the evidence certainly suggests an association. Affective characteristics studied in relation to iron deficiency include irritability, anger, or mood; depression, both as postpartum depression (PPD) or depression independently; and perceived QOL. Differences in assessment tools as well as length and dosage of iron treatment likely play a pivotal role in discordant results. Most studies also include fatigue as a primary outcome as it is closely tied to these affective characteristics.

The aim of this study is to further investigate iron status and iron deficiency symptoms in menstruating females. It builds on the existing research for use of cutoff values for various biochemical assessments of iron as well as for stages of deficiency in which symptoms are experienced. In addition, the association between iron status, measured either biochemically or by self-reported iron deficiency symptoms, and depression was examined.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant
* female
* 18-45 years of age

Exclusion Criteria:

* pregnancy
* male
* outside age range
* post-menopausal
* experiencing one of the following inflammatory or iron metabolism disorders: active treatment for cancer, irritable bowel syndrome, colitis, Chron's disease, chronic heart failure, chronic kidney disease, chronic parasitic infection, hemochromatosis, human immunodeficiency virus, polycystic ovarian syndrome, respiratory illness, sickle cell anemia, and thalassemia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pre-menopausal females
Study Population: Because menstruation causes much lower iron stores in adult females, this study targeted adult, menstruating, non-pregnant females. Additionally, inflammation and iron metabolism disorders can result in biochemical iron values that are difficult to interpret, so these conditions were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
iron deficiency symptoms | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gallaher, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota - Department of Food Science and Nutrition, Saint Paul, Minnesota, United States

DOCUMENTS (3):
  • Study Protocol (2014-01-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT03228173/Prot_000.pdf
  • Informed Consent Form (2015-04-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03228173/ICF_001.pdf
  • Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03228173/SAP_002.pdf